CLINICAL TRIAL: NCT01498757
Title: Genome-wide Association Study to Predict Treatment Response for Chemotherapy in Esophageal Squamous Cell Carcinoma
Brief Title: Genome-wide Association Study
Status: Withdrawn | Type: Observational
Why Stopped: Registration poor
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, Professor of Medicine, Sungkyunkwan University School of Medicine, Department of Hematology and Oncology, Samsung Medical Center
Other Study IDs: 2011-05-076
Record Dates: First submitted 2011-12-21; First posted 2011-12-23 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients treated with Taxane/5-FU/platinum based chemo.

SUMMARY:
To explore biomarkers predictive of clinical response to Taxane/5-FU/platinum based chemotherapy in esophageal squamous cell carcinoma. To identify negative predictive markers to 5-FU/platinum/Taxane. To elucidate signal transduction pathway attributable to 5-FU/platinum/Taxane resistance. To analyze correlation between the quantity of circulating tumor cells and circulating endothelial cell precursors and treatment response to Taxane/5-FU/platinum based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmed esophageal squamous cell carcinoma
* Patients treated with Taxane or 5-FU or platinum based chemotherapy.
* provision of a signed written informed consent.

Exclusion Criteria:

* patients not signed written informed consent.
* patient unacceptable for study in the judgement of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Esophageal squamous cell carcinoma Patients treated with Taxane/5-FU/platinum based chemotherapy.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2012-07-03 (Actual)

PRIMARY OUTCOMES:
Biomarkers predictive | 24months
  Biomarkers predictive of clinical response to Taxane or 5-fluorouracil or platinum based chemotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung medical Center, Seoul, South Korea